CLINICAL TRIAL: NCT03114891
Title: Accelerated TMS to a Novel Brain Target in MDD and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 826007
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Post Traumatic Stress Disorder; Major Depressive Disorder
Keywords: post-traumatic stress; depression; ptsd; tms
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation; potassium channel subfamily K member 3

STUDY DESIGN:
Intervention Model Description: This is a randomized study. All subjects will receive active TMS, so there is no placebo or sham condition. However, the patients will be blinded as to whether or not their site of stimulation is based on the standard targeting method or our novel fMRI-guided targeting method. TMS is administered over to one of these two sites over a two week period, and then TMS will be administered to the other site over a subsequent two-week period. All subjects will receive TMS to both sites as a part of the study, but the order is randomized and counterbalanced.
Who Masked: Participant, Care Provider
Masking Description: The patients will be blinded as to whether or not their site of stimulation is based on the standard targeting method or our novel fMRI-guided targeting method. In addition, staff members administering TMS will not know if the site of stimulation was created based on the standard targeting method or novel fMRI method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- First Round: fMRI-guided Target/Video, Second Round: 6cm Target/Task (Experimental): First round: This site of stimulation will be created from participants' individualized resting connectivity data. We will identify a cortical target in the left prefrontal cortex (LPFC) that influences the subgenual anterior cingulate cortex (sgACC). Two daily sessions (~10min apart) of intermittent theta-burst stimulation will be administered to this fMRI-guided target for 10 consecutive weekdays. Between the two iTBS sessions, participants will watch a relaxing nature video.
  Second round: After 3 weeks, participants will undergo another set of two daily iTBS sessions for 10 consecutive weekdays to their 'standard' target (6cm anterior of their hand knob). Between the two iTBS sessions, participants will complete a working memory task.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Behavioral: Task; Procedure: fMRI-guided TMS target
- First Round: 6cm Target/Video, Second Round: fMRI-guided Target/Task (Experimental): First round: This 'standard' target will be identified by measuring 6cm anterior of the hand knob. Two daily sessions (~10min apart) of intermittent theta-burst stimulation will be administered to this to this target for 10 consecutive weekdays. Between the two iTBS sessions, participants will watch a relaxing nature video.
  Second round: After 3 weeks, participants will undergo another set of two daily iTBS sessions for 10 consecutive weekdays to their fMRI-guided target (cortical target influencing sgACC). Between the two iTBS sessions, participants will complete a working memory task.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Behavioral: Task; Procedure: fMRI-guided TMS target
- First Round: fMRI-guided Target/Task, Second Round: 6cm Target/Video (Experimental): First round: This site of stimulation will be created from participants' individualized resting connectivity data. We will identify a cortical target in the left prefrontal cortex (LPFC) that influences the subgenual anterior cingulate cortex (sgACC). Two daily sessions (~10min apart) of intermittent theta-burst stimulation will be administered to this fMRI-guided target for 10 consecutive weekdays. Between the two iTBS sessions, participants will complete a working memory task.
  Second round: After 3 weeks, participants will undergo another set of two daily iTBS sessions for 10 consecutive weekdays to their 'standard' target (6cm anterior of their hand knob). Between the two iTBS sessions, participants will watch a relaxing nature video.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Behavioral: Task; Procedure: fMRI-guided TMS target
- First Round: 6cm Target/Task, Second Round: fMRI-guided Target/Task (Experimental): First round: This 'standard' target will be identified by measuring 6cm anterior of the hand knob. Two daily sessions (~10min apart) of intermittent theta-burst stimulation will be administered to this to this target for 10 consecutive weekdays. Between the two iTBS sessions, participants will complete a working memory task.
  Second round: After 3 weeks, participants will undergo another set of two daily iTBS sessions for 10 consecutive weekdays to their fMRI-guided target (cortical target influencing sgACC). Between the two iTBS sessions, participants will watch a relaxing nature video.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Behavioral: Task; Procedure: fMRI-guided TMS target

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial Magnetic Stimulation (TMS) is a non-invasive form of brain stimulation. TMS can influence activity in various brain regions, and it allows researchers to test or modify brain circuit communication. In this study, we used administered theta burst TMS stimulation.
Behavioral: Task — Subject completes a working memory task (Letter Nback) between the two rounds of theta burst stimulation.
Procedure: fMRI-guided TMS target — Administration of TMS to individualized targeting from the participant's fMRI scans. Our preliminary data suggest this target region is particularly effective at influencing the sgACC.

SUMMARY:
This is a Clinical Trial designed to evaluate novel transcranial magnetic stimulation (TMS) methods for treating depression/PTSD. TMS is an FDA-approved procedure for treatment-resistant depression. The use of the stimulation in this current study is considered experimental. The purpose of this research study is to compare the effects of TMS at two different brain regions. This information will help the investigators to determine which treatment strategies provide the greatest clinical benefit to patients. Results of the study will provide brain and behavior measures for future work, which may be critical to developing effective disease markers and novel treatments for psychiatric conditions.

DETAILED DESCRIPTION:
Non-invasive transcranial magnetic stimulation (TMS) is now FDA-approved for the treatment of major depressive disorder (MDD). However, there is growing evidence that the targeting strategy for delivering TMS treatment would yield superior clinical outcomes if it were more tailored to individual neuroanatomy. The current study take this idea one step further and suggest that functional MRI guided TMS might yield an even greater leap forward in promoting optimal clinical outcomes.

The sgACC has been well established as a brain area sensitive to negative mood inductions and implicated in neural abnormalities associated with affective and stress disorders. It is therefore one of the primary targets for deep brain stimulation (DBS) treatment of MDD using surgically implanted DBS devices. Recent posthoc imaging studies of patients who have undergone TMS treatment for depression suggest that treatment outcomes tended to be better when patients were by chance stimulated in an area of lateral prefrontal cortex that had high levels of functional connectivity with sgACC. Based on this finding and on interleaved TMS/fMRI probe data, the investigators contend that targeting delivery of TMS to the brain surface non-invasively as indicated by sgACC resting functional connectivity may be especially effective in downregulating sgACC and thereby producing superior clinical outcomes.

Researchers have used TMS/fMRI to better understand causal communication among circuits typically examined with resting fMRI alone. Recent work suggests that there are specific sites that, when stimulated, influence subcortical brain areas implicated in affective disorders such as the sgACC. Previously, TMS targets were based on brain atlases mapped onto individual brain surfaces. This proposal will utilize more individualized targeting from participants' own resting connectivity data to guide stimulation that we show is especially effective in influencing downstream brain areas of interest. The investigators will focus on a target region of the lateral prefrontal cortex (LPFC) that data suggest is particularly effective at influencing the sgACC. As an alternative brain target, we will also test the efficacy of the dorsolateral prefrontal cortex as a target given its precedence in the literature as an effective stimulation site for remediating depressive symptoms. The target will be chosen based on an atlas and will adjust the target coordinates based on the inverse of a nonlinear normalization of each participant's brain to standard brain space. Thus, individual anatomical differences will be taken account with this target though without guidance from individual functional imaging data.

To increase generalizability to other disorders and to patients with comorbid anxiety and depression (the typical clinical profile), the investigators will recruit patients who are diagnosed PTSD and have symptoms of depression or those who experience trauma-induced MDD. Participants will be scanned in an MRI to get anatomical and resting fMRI data to guide TMS, then participants will be invited to participate in two rounds of two week TMS treatment to each site (order counterbalanced) with one month between treatments. Participants will be monitored to assess PTSD symptoms, depressive symptoms,and quality of life before, acutely after, and one month following TMS treatments to evaluate the effectiveness of each site in mitigating symptoms or improving functioning.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old, male or female, any race
2. Patients must currently meet sufficient DSM criteria for PTSD and have symptoms of depression; or meet criteria for trauma-induced MDD
3. Capacity to give informed consent and follow study procedures
4. English speaking

Exclusion Criteria:

1. Outside age range
2. Patient does not meet sufficient DSM criteria for PTSD or MDD
3. Psychiatric medication use
4. Significant handicaps (e.g. mental handicap) that would interfere with testing procedures
5. MRI contraindications
6. Additional TMS contraindications
7. Medication use that substantially reduces seizure threshold to TMS (olanzapine, chlorpromazine, lithium)
8. Opiate medication
9. Known neurological disorders including multiple sclerosis, encephalopathy, seizure disorder, brain tumors
10. Current alcohol or substance abuse disorder (moderate or severe)
11. Current schizophrenia or other psychotic disorder, or current bipolar disorder
12. Refusal to abstain from illicit drug use for the duration of the study
13. Refusal to abstain from alcohol within 24 hours of the MRI scan
14. Pregnancy
15. Newly initiated psychotherapy (less than 6 weeks)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Oathes, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen AC, Oathes DJ, Chang C, Bradley T, Zhou ZW, Williams LM, Glover GH, Deisseroth K, Etkin A. Causal interactions between fronto-parietal central executive and default-mode networks in humans. Proc Natl Acad Sci U S A. 2013 Dec 3;110(49):19944-9. doi: 10.1073/pnas.1311772110. Epub 2013 Nov 18. PMID 24248372
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 87 subjects screened for the study, 37 did not start treatment (19 were deemed ineligible,15 withdrew, 3 lost to follow up) and 50 enrolled in the study (assigned to an intervention group).
Groups:
- First Round: 6cm Target/Task, Second Round: fMRI-guided Target/Video: First round: This 'standard' target will be identified by measuring 6cm anterior of the hand knob. Two daily sessions (~10min apart) of intermittent theta-burst stimulation will be administered to this to this target for 10 consecutive weekdays. Between the two iTBS sessions, participants will complete a working memory task.
  Second round: After 3 weeks, participants will undergo another set of two daily iTBS sessions for 10 consecutive weekdays to their fMRI-guided target (cortical target influencing sgACC). Between the two iTBS sessions, participants will watch a relaxing nature video.
Period: First Treatment Round
Arm/Group | First Round: fMRI-guided Target/Video, Second Round: 6cm Target/Task | First Round: 6cm Target/Video, Second Round: fMRI-guided Target/Task | First Round: fMRI-guided Target/Task, Second Round: 6cm Target/Video | First Round: 6cm Target/Task, Second Round: fMRI-guided Target/Video
Started | 12 | 14 | 11 | 13
Completed | 12 | 11 | 10 | 12
Not Completed | 0 | 3 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1
Period: 3 Week Break
Arm/Group | First Round: fMRI-guided Target/Video, Second Round: 6cm Target/Task | First Round: 6cm Target/Video, Second Round: fMRI-guided Target/Task | First Round: fMRI-guided Target/Task, Second Round: 6cm Target/Video | First Round: 6cm Target/Task, Second Round: fMRI-guided Target/Video
Started | 12 | 11 | 10 | 12
Completed | 11 | 10 | 10 | 11
Not Completed | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Second Treatment Round
Arm/Group | First Round: fMRI-guided Target/Video, Second Round: 6cm Target/Task | First Round: 6cm Target/Video, Second Round: fMRI-guided Target/Task | First Round: fMRI-guided Target/Task, Second Round: 6cm Target/Video | First Round: 6cm Target/Task, Second Round: fMRI-guided Target/Video
Started | 11 | 10 | 10 | 11
Completed | 9 | 10 | 10 | 11
Not Completed | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- First Round: fMRI-guided Target/Video: First round: This site of stimulation will be created from participants' individualized resting connectivity data. We will identify a cortical target in the left prefrontal cortex (LPFC) that influences the subgenual anterior cingulate cortex (sgACC). Two daily sessions (~10min apart) of intermittent theta-burst stimulation will be administered to this fMRI-guided target for 10 consecutive weekdays. Between the two iTBS sessions, participants will watch a relaxing nature video.
  Second round: After 3 weeks, participants will undergo another set of two daily iTBS sessions for 10 consecutive weekdays to their 'standard' target (6cm anterior of their hand knob). Between the two iTBS sessions, participants will complete a working memory task.
- First Round: 6cm Target/Video: First round: This 'standard' target will be identified by measuring 6cm anterior of the hand knob. Two daily sessions (~10min apart) of intermittent theta-burst stimulation will be administered to this to this target for 10 consecutive weekdays. Between the two iTBS sessions, participants will watch a relaxing nature video.
  Second round: After 3 weeks, participants will undergo another set of two daily iTBS sessions for 10 consecutive weekdays to their fMRI-guided target (cortical target influencing sgACC). Between the two iTBS sessions, participants will complete a working memory task.
- First Round: fMRI-guided Target/Task: First round: This site of stimulation will be created from participants' individualized resting connectivity data. We will identify a cortical target in the left prefrontal cortex (LPFC) that influences the subgenual anterior cingulate cortex (sgACC). Two daily sessions (~10min apart) of intermittent theta-burst stimulation will be administered to this fMRI-guided target for 10 consecutive weekdays. Between the two iTBS sessions, participants will complete a working memory task.
  Second round: After 3 weeks, participants will undergo another set of two daily iTBS sessions for 10 consecutive weekdays to their 'standard' target (6cm anterior of their hand knob). Between the two iTBS sessions, participants will watch a relaxing nature video.
- First Round: 6cm Target/Task: First round: This 'standard' target will be identified by measuring 6cm anterior of the hand knob. Two daily sessions (~10min apart) of intermittent theta-burst stimulation will be administered to this to this target for 10 consecutive weekdays. Between the two iTBS sessions, participants will complete a working memory task.
  Second round: After 3 weeks, participants will undergo another set of two daily iTBS sessions for 10 consecutive weekdays to their fMRI-guided target (cortical target influencing sgACC). Between the two iTBS sessions, participants will watch a relaxing nature video.
- Total: Total of all reporting groups
Arm/Group | First Round: fMRI-guided Target/Video | First Round: 6cm Target/Video | First Round: fMRI-guided Target/Task | First Round: 6cm Target/Task | Total
Number analyzed (Participants) | 12 | 14 | 11 | 13 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 11 | 13 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.25 (13.79) | 36.42 (12.06) | 29.27 (8.45) | 36 (10.56) | 34.46 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 8 | 8 | 31
  Male | 4 | 7 | 3 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 1 | 5
  Not Hispanic or Latino | 11 | 12 | 8 | 11 | 42
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 1 | 7
  White | 8 | 8 | 5 | 9 | 30
  More than one race | 1 | 1 | 2 | 2 | 6
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 4
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire(PHQ)-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression.
  The scale has nine items, each of which is scored 0 to 3, providing a 0 to 27 severity score. Higher score represents worse outcome. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
  units on a scale | 15.08 (5.21) | 15.43 (4.69) | 16 (4.77) | 17.85 (3.21) | 16.10 (4.51)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Depression Severity of TMS at fMRI-guided Brain Target vs Standard Brain Target
Description: We used the Montgomery-Asberg Depression Rating Scale (MADRS) to measure depression severity after TMS at fMRI-guided brain target vs standard brain target. The MADRS is clinician-rated and consists of 10 items; each item is rated on a 0-6 scale, resulting in a maximum total score of 60 points. Higher MADRS score indicates more severe depression.
  For this outcome, we calculated the change (percent decrease) from the participant's baseline MADRS score to their MADRS score after the first round of TMS (to either fMRI-guided brain target or standard brain target). If the outcome is positive, there was a reduction in the MADRS total score, or a reduction in the presence of depressive symptoms after TMS. If the change is negative, there was an increase in the MADRS total score, or an increase in the presence of depressive symptoms after TMS.
  Higher positive values means better outcome (or more symptom reduction).
Time Frame: Before and after the first round of two weeks of TMS treatment (two daily iTBS sessions over 10 consecutive weekdays)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | First Round: fMRI-guided Target/Video, Second Round: 6cm Target/Task | First Round: 6cm Target/Video, Second Round: fMRI-guided Target/Task | First Round: fMRI-guided Target/Task, Second Round: 6cm Target/Video | First Round: 6cm Target/Task, Second Round: fMRI-guided Target/Task
Number analyzed (Participants) | 12 | 11 | 10 | 12
percentage of change | 49.11 (25.42) | 24.94 (37.97) | 36.47 (33.91) | 42.56 (30.75)

ADVERSE EVENTS:
Time Frame: Up to 2 weeks for each intervention
Description: Safety population included all participants who received at the one round of TMS intervention.
  Our adverse event definition includes all the specifications of the clinicaltrials.gov definition, but it also includes 'any symptom, sign, illness or experience that the Principal Investigator determines as significantly worse during course of the study'. Thus, our definition considers non-medical occurrences as AEs.
Groups:
- fMRI-guided Target/Video: Two daily rounds (~10min apart) of intermittent theta-burst stimulation to the fMRI-guided target for 10 consecutive weekdays. Between the two rounds of TMS, participants watched a relaxing nature video.
- 6cm Target/Video: Two daily rounds (~10min apart) of intermittent theta-burst stimulation to the 'standard' or 6cm target for 10 consecutive weekdays. Between the two rounds of TMS, participants watched a relaxing nature video.
- fMRI-guided Target/Task: Two daily rounds (~10min apart) of intermittent theta-burst stimulation to the fMRI-guided target for 10 consecutive weekdays. Between the two iTBS sessions, participants will complete a working memory task.
- 6cm Target/Task: Two daily rounds (~10min apart) of intermittent theta-burst stimulation to the 'standard' or 6cm target for 10 consecutive weekdays. Between the two iTBS sessions, participants will complete a working memory task.
Arm/Group | fMRI-guided Target/Video | 6cm Target/Video | fMRI-guided Target/Task | 6cm Target/Task
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24 | 0/21 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 7/24 | 2/21 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | fMRI-guided Target/Video (N=23) | 6cm Target/Video (N=24) | fMRI-guided Target/Task (N=21) | 6cm Target/Task (N=24)
Headache (General disorders) | 0 (0) | 4 (13) | 2 (3) | 0 (0) — TMS-induced headache.
Scalp muscle/Facial muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Muscle tenderness or pain in scalp and/or facial muscles during/after TMS stimulation.
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) — Jaw pain from TMS muscle activation.
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant developed and was diagnosed with Bell's Palsy during first six days of TMS treatment. It was determined this was unrelated to study procedures.
Dizziness and disorientation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Dizziness and disorientation after TMS administration.
Worsening of symptoms (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) — Subjects reported increase in anxiety and suicidal symptoms/behaviors during their study participation. PI determined this was unrelated to study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT03114891/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03114891/ICF_001.pdf